CLINICAL TRIAL: NCT02884115
Title: Randomized, Clinical Trial to Compare the Serological Response Rates of Serofast Early Syphilis Cases Retreated With Three Doses Benzathine Penicillin and Absence of Any Retreatment
Brief Title: Serological Response to Retreatment of Serofast Early Syphilis Cases With Benzathine Penicillin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Jun Li, M.D., Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-2016080
Record Dates: First submitted 2016-08-22; First posted 2016-08-30 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Syphilis
MeSH Terms: conditions — Syphilis | interventions — Penicillin G Benzathine

ARMS (2):
- Retreatment group (Active Comparator): Serofast early syphilis cases retreated with three doses benzathine penicillin
  Interventions: Drug: benzathine penicillin
- Control group (No Intervention): Absence of any retreatment

INTERVENTIONS:
Drug: benzathine penicillin
  Arms: Retreatment group

SUMMARY:
A continuing challenge to determining the response to treatment of early syphilis (primary, secondary, early latent syphilis) is exemplified by the substantial proportion of patients who fail to achieve serological cure and remain serofast. Although retreatment is often done in clinical practice, optimal management remains uncertain due to the paucity of data regarding serological response to retreatment and long-term outcomes. Furthermore, the investigators cannot rule out that the gradually increasing seroreversion/serological cure rates may have been due to the natural decline in rapid plasma regain (RPR) titers after initial therapy, rather than due to the additional dose of benzathine penicillin. Thus, the investigators would like to conduct a clinical trial to compare the serological response rates of serofast early syphilis cases retreated with three doses benzathine penicillin and absence of any retreatment (control group).

ELIGIBILITY:
Inclusion Criteria:

* Early Syphilis Cases Determined to Be Serofast at 6 Months after Initial Treatment

Exclusion Criteria:

* Human immunodeficiency virus (HIV)-infected
* Baseline serology showed a nonreactive RPR test
* follow-up is inadequate
* Allergic to penicillin
* Pregnant woman

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-08; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Rapid plasma regain titer | 6 months after retreatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology and Venereology, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China, Beijing, China